CLINICAL TRIAL: NCT05384834
Title: Incorporating Cardiovascular Risk Assessment Into Adolescent and Young Adult Visits to Improve Cardiovascular Health
Brief Title: Incorporating CV Risk Assessment in AYA Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Holly Gooding, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001418; 1R03HL155253-01 (NIH)
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA participants (Experimental): AYA participants will complete a brief initial survey consisting of demographic information and the Visual Analog Scale (VAS) and the #HerHeart tool in clinic. AYA participants will the rate the usability of the #HerHeart tool using the Website Analysis and Measurement Inventory (WAMMI), the likelihood they would recommend the app to their friends, and the likelihood of behavior change. AYA participants will then be offered the opportunity to continue into the 3-month intervention phase.
  Interventions: Behavioral: #HerHeart tool

INTERVENTIONS:
Behavioral: #HerHeart tool — An integrated application consisting of a lifestyle-based CVD risk assessment and companion behavioral intervention. It will be administered at baseline and 3 months follow-up.

SUMMARY:
The purpose of this study is to evaluate the web tool #HerHeart's usability and feasibility in adolescent and young adult women (AYA) and the opinion of their healthcare providers (HCP).

DETAILED DESCRIPTION:
The objective of the proposed research is to increase young women's perceived susceptibility to CVD and provide a cue to action to adopt heart-healthy behaviors. The aim of the proposed study is to evaluate the usability and initial feasibility of #HerHeart. The investigators will recruit 30 AYA participants and will ask 10 HCPs to evaluate the usability and feasibility of the web tool.

The study population will include female patients ages 13-21 years from the CHOA Adolescent Medicine Practice and Grady Teen Health Program. Part of our study population will be considered vulnerable (children under the age of 18 years). Subjects will be recruited via phone in advance of a clinical visit, from the waiting rooms of each clinic at the time of their appointment (in-person) or via Zoom at a time scheduled after their telehealth appointment (virtual). Written informed consent will be obtained for subjects 18 years and older. For subjects younger than 18 years, written parental permission (unless doing so would violate the adolescents' right to privacy, in which the Waiver of Parental Permission will be invoked) and written informed assent will be obtained. All consent procedures will take place in a private research room of each clinic (for in-person visits) or via Zoom videoconferencing (for virtual visits). Participants who agree to participate will attend a study visit at the Emory Children's Center Research Unit.

Data for this study will be collected from participants via surveys/questionnaires, and semi-structured interviews that will be audio-recorded. Data collected will include demographic information, cardiovascular disease risk information, health metrics (BMI, blood pressure), cognitive data (perceived stress, quality of life), and participant feedback on a mobile app intervention. All subjects will receive a study identification number. Only the PI will have the codes linking the study identification numbers to subjects and these codes will be stored in a locked cabinet. All data will be collected in a private research room in the clinics (in-person visits) or in a password-protected Zoom videoconference (virtual). All study staff will complete biomedical or socio-behavioral training through the Collaborative IRB Training Initiative Program (CITI). Data will be stored on the Emory servers in password-protected files.

ELIGIBILITY:
Inclusion Criteria (AYAs):

* Patient at CHOA Hughes Spalding Adolescent Medicine Practice or the Grady Health System Teen Program
* Age 13-21 years
* Self-identifying as non-Hispanic Black or White race (inclusive of Hispanic ethnicity)
* Self-identifying as female
* Visit type is annual wellness/health check, behavioral/mental health, or reproductive/gynecological health
* Consistent access to a mobile device with internet capability

Exclusion Criteria (AYAs):

* Cognitive impairment limiting ability to complete study procedure
* Spoken and written language other than English
* Diagnosis of hypertension, diabetes, or hyperlipidemia requiring medications, or atherosclerotic cardiovascular disease
* Past or current diagnosis of a DSM-V eating disorder
* Diagnosis of schizophrenia, bipolar disorder, or psychiatric hospitalization in the past 12 months
* Pregnant at the time of the study.

Inclusion Criteria (HCPs) to complete feasibility surveys:

* Clinical team member (physician or nurse practitioner, nurse, social worker, psychologist, health educator, medical assistant, dietitian) at the CHOA Hughes Spalding Adolescent Medicine Practice or the Grady Health System Teen Program
* Practicing at one of the study sites at least twice per month on average over the past year

Exclusion Criteria (HCPs)

* Member of the research study team

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Gooding, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta - Hughes Spalding Research Room, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Children's Healthcare of Atlanta - Hughes Spalding Research Room in Atlanta, Georgia, USA. Participant enrollment began July 01, 2022, and all follow-up assessments were completed by April 03, 2023.
Pre-assignment Details: The healthcare providers (HCPs) were instructed to complete a short anonymous survey without demographic information. Demographic information was not required to answer the survey. HCPs were not enrolled. They were not actually part of the clinical trial, per the NIH definition of a clinical trial.
Period: Overall Study
Arm/Group | AYA Participants
Started | 60
Completed | 12
Not Completed | 48
Not completed — Lost to Follow-up | 43
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All participants who provided consent to participate in the study
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 17 [13 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 50
  White | 1
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: #HerHEART Risk Score in AYA From Baseline
Description: Risk is assessed based on answers surrounding the most critical diet and lifestyle factors that can influence a person's CVD risk. The factors include exercise, intake of fruits, vegetables, grains, nuts, sugary beverages and red/processed meats, and exercise. The Healthy Heart Score algorithm will be used to calculate the relative percent risk score of participants. Participants with a higher percent risk score have a higher risk for CVD based on their current reported habits. Those at low risk will have a risk score <10%, moderate risk a risk score between 10 and 15%, and high risk a score above 15%.
Time Frame: Baseline, 3 months post-enrollment
Population: Includes all participants who completed the baseline questionnaires, and the three months follow-up includes only those who completed the study activities at the specific time point. Even though twelve (12) participants completed all activities, data was lost on 2 individuals. HCPs, n=5 from the same two clinical practices in Atlanta, Georgia were recruited by the research coordinator only to understand their perspectives about incorporating the HerHeart tool into clinical practice.
Measure: Median (Inter-Quartile Range); unit: Percentage Risk
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Percentage Risk
  Baseline | 0.10 [0.07 to 0.13]
  Three (3) months post-enrollment: number analyzed (Participants) | 10
  Three (3) months post-enrollment | 0.08 [0.06 to 0.10]

2. Primary Outcome: Overall Composite of Diet Score
Description: Diet score = (0.03626 × grams/d of cereal fiber + 0.18283 [if fruits + vegetables ≥3 servings/d] + 0.14522 [if nuts 0.1-1 servings/d + 0.2444 [if nuts >1 servings/d]- 0.14631 × servings/d of sugar-sweetened beverages - 0.15624 × servings/d of red and processed meats)*10 A higher score implies better diet quality. An increase in diet score correlates with a better outcome.
Time Frame: Baseline, 3 months months post-enrollment
Population: Includes all participants who completed the baseline questionnaires, and the three-month follow-up includes only those who completed the study activities at the specific time point. Even though twelve (12) participants completed all activities, data was lost on 2 individuals.
Measure: Median (Inter-Quartile Range); unit: Diet Score
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Diet Score
  Baseline | 0.27 [-0.84 to 1.11]
  Three (3) months post-enrollment: number analyzed (Participants) | 10
  Three (3) months post-enrollment | 0.28 [-0.84 to 1.11]

3. Primary Outcome: Fruit and Vegetable Intake
Description: Intake will be measured with number of servings per day. Increase in servings/day correlates with a better outcome.
Time Frame: Baseline, 3 months post- post-enrollment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Number of Servings per day
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Number of Servings per day
  Fruits at Baseline | 2.00 [1.00 to 3.00]
  Fruits at 3 months post-enrollment: number analyzed (Participants) | 10
  Fruits at 3 months post-enrollment | 1.5 [1.00 to 3.00]
  Vegetables at Baseline | 1.00 [0.88 to 2.00]
  Vegetables at 3 months post-enrollment: number analyzed (Participants) | 10
  Vegetables at 3 months post-enrollment | 2.00 [1.00 to 2.00]

4. Primary Outcome: Red and Processed Meats Intake
Description: Intake will be measured with number of servings per day. A decrease in consumption is associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: number of servings per week
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
number of servings per week
  Red meats at baseline | 0.30 [0.30 to 0.50]
  Red meats at 3 months post-enrollment: number analyzed (Participants) | 10
  Red meats at 3 months post-enrollment | 0.30 [0.30 to 0.88]
  Processed Meats at Baseline | 0.50 [0.30 to 1.00]
  Processed Meats at 3 months post-enrollment: number analyzed (Participants) | 10
  Processed Meats at 3 months post-enrollment | 0.30 [0.10 to 0.45]

5. Primary Outcome: Sugar and Sweetened Beverages
Description: Intake will be measured with number of servings per week. A decrease in consumption is associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: number of servings per week.
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
number of servings per week.
  Baseline | 0.30 [0.10 to 0.50]
  Three months post-enrollment: number analyzed (Participants) | 10
  Three months post-enrollment | 0.30 [0.15 to 0.45]

6. Primary Outcome: Nut Consumption
Description: Intake will be measured with number of servings per week. An increase in intake is associated with a better outcome.
Time Frame: Baseline, 3 months post-intervention
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Number of Servings per week
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Number of Servings per week
  Baseline | 0.30 [0.00 to 0.30]
  3 months post-intervention: number analyzed (Participants) | 10
  3 months post-intervention | 0.30 [0.15 to 0.45]

7. Primary Outcome: Alcohol Consumption
Description: Number of participants who consume alcohol will be collected. No alcohol consumption is associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Participants
  Baseline | 0
  3 months post-enrollment: number analyzed (Participants) | 10
  3 months post-enrollment | 0

8. Primary Outcome: Nicotine Use
Description: Self-reported smoker status will be obtained and classified as: Never smoke, used to smoke, current smoker. Investigators will look at changes in smoking status where a decrease in use is associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
Participants
  Baseline: Never Smoke | 46
  Baseline: Used to Smoke | 4
  Baseline: Current Smoker | 10
  Three months post-enrollment: number analyzed (Participants) | 10
  Three months post-enrollment: Never Smoke | 9
  Three months post-enrollment: Used to Smoke | 1
  Three months post-enrollment: Current Smoker | 0

9. Primary Outcome: Cereal Fiber
Description: Consumption of cereal will be measured in g/day. An increase in cereal fiber is associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: g/day
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
g/day
  Baseline | 0.30 [0.30 to 0.50]
  Three months post-enrollment: number analyzed (Participants) | 10
  Three months post-enrollment | 0.30 [0.30 to 0.50]

10. Primary Outcome: Physical Activity
Description: Physical activity will be measured in number of hours per week. Increase in physical activity associated with a better outcome.
Time Frame: Baseline, 3 months post-enrollment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: number of hours per week
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
number of hours per week
  Intense Physical Activity at Baseline | 0.75 [0.00 to 1.06]
  Intense Physical Activity at 3 months post-enrollment: number analyzed (Participants) | 10
  Intense Physical Activity at 3 months post-enrollment | 0.75 [0.06 to 2.00]
  Moderate Physical Activity at Baseline | 0.75 [0.63 to 2.00]
  Moderate Physical Activity at 3 months post-enrollment: number analyzed (Participants) | 10
  Moderate Physical Activity at 3 months post-enrollment | 1.38 [0.75 to 2.00]

11. Secondary Outcome: BMI From Baseline
Description: AYA participant's BMI will be measured during the clinic appointment when participant is recruited. AYA participants will then be asked to return for a study visit 3 months post intervention where their BMI will be measured again. Change in BMI will be measured with a decrease in BMI being associated with a positive outcome and an increase in BMI being associated with a negative outcome.
Time Frame: Baseline, 3 month post-enrollment
Population: Includes all participants who completed the baseline questionnaires, and the three months follow-up includes only those who completed the study activities at the specific time point.
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
kg/m^2
  BMI at Baseline | 24 [21 to 28]
  BMI at 3 months post-enrollment: number analyzed (Participants) | 12
  BMI at 3 months post-enrollment | 25 [23 to 25]

12. Secondary Outcome: Systolic Blood Pressure (BP) From Baseline
Description: AYA participants' systolic BP (SBP) will be measured during the clinic appointment when the participant is recruited. AYA participants will then be asked to return for a study visit 3 months post-intervention where their BP will be measured again. Change in SBP will be measured with a decrease in SBP being associated with a positive outcome and an increase in SBP being associated with a negative outcome.
Time Frame: Baseline, 3 month post-enrollment
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
mmHg
  SPB at Baseline | 118 [112 to 121]
  SBP at 3 months post-enrollment: number analyzed (Participants) | 12
  SBP at 3 months post-enrollment | 117 [108 to 133]

13. Secondary Outcome: Diastolic Blood Pressure (BP) From Baseline
Description: AYA participants' diastolic BP (DBP) will be measured during the clinic appointment when the participant is recruited. AYA participants will then be asked to return for a study visit 3 months post-intervention where their BP will be measured again. Change in DBP will be measured with a decrease in diastolic BP being associated with a positive outcome and an increase in BP being associated with a negative outcome.
Time Frame: Baseline, 3 month post-enrollment
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | AYA Participants
Number analyzed (Participants) | 60
mmHg
  Baseline DBP | 67 [63 to 71]
  DBP at 3 months post-enrollment: number analyzed (Participants) | 12
  DBP at 3 months post-enrollment | 67 [62 to 72]

ADVERSE EVENTS:
Time Frame: Data collection from study enrollment until study participation was completed, up to 3 months post-enrollment.
Groups:
- AYA Participants: AYA participants will complete a brief initial survey consisting of demographic information, the Visual Analog Scale (VAS), and the #HerHeart tool in the clinic. AYA participants will rate the usability of the #HerHeart tool using the Website Analysis and Measurement Inventory (WAMMI), the likelihood they would recommend the app to their friends, and the likelihood of behavior change. AYA participants will then be offered the opportunity to continue into the 3-month intervention phase.
  * HerHeart tool: An integrated application consisting of a lifestyle-based CVD risk assessment and companion behavioral intervention. It will be administered at baseline and 3 months follow-up.
Arm/Group | AYA Participants
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05384834/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT05384834/ICF_002.pdf